CLINICAL TRIAL: NCT01202110
Title: A Phase II, Dose Escalation, Single Center Study on the Effects of Early Propranolol on Heart Rate, Blood Pressure, and Cerebral Perfusion Pressure in Subjects Who Present With Moderate to Severe Traumatic Brain Injury.
Brief Title: Early Propranolol After Traumatic Brain Injury: Phase II
Acronym: EPAT: Phase II
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Eric Ley, MD, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00020850
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Experimental): Propranolol 1mg iv
  Interventions: Drug: Propranolol
- Control (No Intervention): Routine care

INTERVENTIONS:
Drug: Propranolol
  Arms: Propranolol

SUMMARY:
The primary objective of this study is to determine in patients with traumatic brain injury (TBI) the safe dosing of propranolol. Safety will be measured by episodes of bradycardia (heart rate < 60 beats per minute), hypotension (defined as systolic blood pressure < 90) or decreased cerebral perfusion pressure (defined as CPP less than 60mmHg) that are refractive to Brain Trauma Foundation guidelines for treatment. A no-treatment arm will establish the number of episodes of bradycardia, hypotension and reduced cerebral pressure refractory to treatment that occur without propranolol.

ELIGIBILITY:
Inclusion Criteria:

* patients who present within 6 hours of traumatic brain injury who have 1) a Glasgow Coma Scale (GCS) score of ≤8 or a GCS of 9-12 with computerized tomography brain scans demonstrating brain injury.

Exclusion Criteria:

* pregnancy,
* patients already treated with beta-blockers,
* patients treated for antiarrhythmic, immunosuppressive or antiinfective treatment,
* myocardial infarction during the last 3 months,
* unstable or severe heart disease,
* severe chronic obstructive pulmonary disease,
* serious liver disease,
* cardiac ischemia that prevents the initiation of vasopressors,
* signs of cardiac arrhythmia or heart block on EKG,
* ischemic limb disease that prevents the initiation of vasopressors, vasopressors at maximum dose defined as norepinephrine at 40µg/min or neosynephrine at 300µg/min.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Control
- Propranolol: Propranolol
Period: Overall Study
Arm/Group | Control | Propranolol
Started | 10 | 0
Completed | 10 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Control
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Determine in Patients With Traumatic Brain Injury (TBI) the Safe Dosing of Early Propranolol.
Description: The primary outcome is to determine the safety of early propranolol treatment after TBI by recording the number of episodes of bradycardia (heart rate < 60 beats per minute), hypotension (defined as systolic blood pressure < 90) or decreased cerebral perfusion pressure (defined as CPP less than 60mmHg) refractive to treatment.
Time Frame: 24 months
Population: Terminated prior to enrolling
Groups:
- Propranolol: 0
Arm/Group | Propranolol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Control: 10
Arm/Group | Control
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes